CLINICAL TRIAL: NCT03200743
Title: Relationship Between Catestatin and Pregnant Hypertensive Disorders
Brief Title: Catestatin and Hypertension in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yuchen Pan (Other)
Responsible Party: Sponsor-Investigator, Yuchen Pan, Peking University Third Hospital, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Other Study IDs: 20170513
Record Dates: First submitted 2017-06-19; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Pre-Eclampsia; Eclampsia; Hypertension, Pregnancy-Induced; Hypertension in Pregnancy
Keywords: Hypertension; Pregnancy; Catestatin
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia; Hypertension, Pregnancy-Induced; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Years
Biospecimen Retention: None Retained — Plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hpertension
- Health

SUMMARY:
Catestatin is a kind of protein involved with cardiovascular disease. Accumulated evidence shows that Catestatin may be a predictor of primary hypertension, but whether it plays the same role in pregnant hypertensive disorders needs to be determined. By measuring the plasma level of Catestatin, main biochemical marks and UCG in healthy pregnancy and pregnancy with hypertension, the research may contribute to this problem.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy women
* Pregnancy women with hypertension

  1. Despite the pregnant gestational age , systolic blood pressure ≥140 mm Hg OR a diastolic blood pressure of ≥90 mm Hg measured three times more than 24 hours apart
  2. Pregnant gestational age > 20 weeks, systolic blood pressure ≥140 mm Hg OR a diastolic blood pressure of ≥90 mm Hg measured twice more than 4 hours apart

Exclusion Criteria:

* Lack of blood sample at the specified enrollment period
* Women who refuse the study
* Other illness which needs medications interfering with blood pressure (eg: Asthma requiring systemic steroids)
* Known coronary artery disease or heart failure
* Serious medical illness (eg: renal insufficiency, congestive heart disease, chronic respiratory insufficiency, uncontrolled infection).
* multiple endocrine neoplasia or Cushing's syndrome or mixed tumours or pheochromocytoma or medullary thyroid carcinoma.
* previous history of malignant tumour, with the exception of carcinoma in situ of the uterine cervix or non-melanoma skin cancer
* renal insufficiency

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in Peking University Third Hospital maternity ward after May, 2017
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-05-14 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
plasma level of Catestatin | once at the specified enrollment period
  plasma level of Catestatin with the unit "mmol/l"

SECONDARY OUTCOMES:
blood pressure | the specified enrollment period,42 days and 2 months after the pregnancy
  systolic and diastolic blood pressure with the unit "mmHg"

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijin, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided